CLINICAL TRIAL: NCT06767280
Title: Tensiomyography Evaluation of Gastrocnemius Muscles in Individuals with Chronic Lumbar Radiculopathy
Brief Title: Tensiomyography of Gastrocnemius in Lumbar Radiculopathy
Acronym: TMGGLR
Status: Recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Mostafa Zaki Nassef, Master's Student, Faculty of Physiotherapy, Cairo University, Cairo University
Other Study IDs: (No: P.T.REC/012/005417)
Record Dates: First submitted 2024-12-31; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Tensiomyography; Gastrocnemius Muscle Assessment; Chronic Lumbar Radiculopathy
Keywords: Chronic Lumbar Radiculopathy; Tensiomyography (TMG); Gastrocnemius Muscles; Neuromuscular Function; Muscle Assessment; Electrophysiology

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Right Leg TMG measurements for the right leg. Left Leg TMG measurements for the left leg.: Right Leg Neuromuscular characteristics of the right leg measured using TMG in patients with chronic lumbar radiculopathy.
  Left Leg Neuromuscular characteristics of the left leg measured using TMG in patients with chronic lumbar radiculopathy.

SUMMARY:
This cross-sectional study aims to evaluate the neuromuscular characteristics of the gastrocnemius muscles in individuals with chronic lumbar radiculopathy using tensiomyography (TMG). By analyzing parameters such as muscle contraction time, displacement, and relaxation time, the study seeks to understand potential alterations in muscle properties that may contribute to functional limitations in this patient population. Findings from this research may provide valuable insights into the role of gastrocnemius muscles in neuromuscular dysfunction and inform tailored rehabilitation strategies.

DETAILED DESCRIPTION:
Lumbar radiculopathy is a condition characterized by the compression or irritation of one or more nerve roots in the lumbar spine, often resulting in pain, weakness, numbness, or difficulty controlling specific muscles. The primary causes of lumbar radiculopathy include herniated discs, spinal stenosis, and degenerative disc disease. These conditions lead to nerve root compression, resulting in radiating pain down the leg, commonly referred to as sciatica.

The impact of lumbar radiculopathy extends beyond pain, affecting muscle function and neuromuscular control. The involvement of nerve roots such as L4, L5, and S1 can particularly affect the muscles in the lower extremities, including the plantar flexor muscles, which are crucial for movements like walking, running, and maintaining balance. These muscles, namely the gastrocnemius and soleus, play a pivotal role in plantar flexion, an essential motion for locomotion.

In individuals with lumbar radiculopathy, the neural input to these muscles can be compromised, leading to muscle weakness, altered reflexes, and changes in muscle activation patterns. Studies have shown that patients with lumbar radiculopathy often exhibit decreased muscle strength and endurance in the affected lower extremity. These neuromuscular deficits can contribute to impaired gait mechanics and an increased risk of falls, significantly affecting the quality of life.

Tensiomyography (TMG) is a non-invasive diagnostic tool used to assess the contractile properties of skeletal muscles. TMG measures the muscle belly's displacement in response to a standardized electrical stimulus, providing valuable information about muscle function. Key parameters measured by TMG include contraction time (Tc), delay time (Td), sustain time (Ts), relaxation time (Tr) and Displacement (Dm) reflecting the muscle's response speed, duration of contraction, and recovery.

TMG has gained popularity in both clinical and sports settings due to its ability to detect muscle imbalances, monitor rehabilitation progress, and guide training programs. Its non-invasive nature and the detailed information it provides make it an ideal tool for assessing muscle health and function in various populations, including those with neuromuscular disorders.

The intersection of lumbar radiculopathy, plantar flexor muscle function, and TMG presents a compelling area of study. The nerve root compression in lumbar radiculopathy can lead to altered neuromuscular control of the plantar flexor muscles, resulting in changes in muscle contractile properties. TMG can effectively capture these changes, providing insights into the extent of neuromuscular impairment and guiding targeted rehabilitation strategies.

Studies utilizing TMG have demonstrated significant differences in the contractile properties of muscles in individuals with lumbar radiculopathy compared to healthy controls. For instance, longer contraction and relaxation times in the plantar flexor muscles indicate a delay in muscle response and recovery, which could be attributed to compromised neural input from the affected lumbar nerve roots. These findings underscore the importance of neuromuscular assessments in patients with lumbar radiculopathy.

By identifying specific deficits in muscle function, TMG can help clinicians design individualized rehabilitation programs aimed at restoring normal muscle activity and improving overall functional outcomes. Rehabilitation strategies may include strength training, neuromuscular re-education, and proprioceptive exercises tailored to address the specific impairments identified through TMG assessments.

Recent research has focused on the application of TMG in various clinical settings, including the assessment of neuromuscular disorders like lumbar radiculopathy. These studies provide evidence supporting the use of TMG as a reliable tool for evaluating muscle function and guiding rehabilitation.

The integration of TMG in evaluating the plantar flexor muscles in individuals with chronic lumbar radiculopathy provides a nuanced understanding of the neuromuscular impairments associated with this condition. By leveraging the detailed insights from TMG assessments, clinicians can develop targeted rehabilitation strategies to improve muscle function, enhance mobility, and ultimately, the quality of life for patients suffering from lumbar radiculopathy. The ongoing research and clinical applications of TMG continue to expand its utility, offering promising avenues for advancing neuromuscular diagnostics and rehabilitation

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-55 years.
* Clinical diagnosis of chronic lumbar radiculopathy confirmed by MRI and clinical examination.
* Presence of symptoms for more than 12 weeks.
* One limb is affected by the condition, while the other limb is unaffected and will serve as the control.

Exclusion Criteria:

* ● Acute lumbar radiculopathy (symptoms less than 12 weeks).

  * History of lower limb surgery or severe musculoskeletal disorders affecting the plantar flexor muscles.
  * Neurological disorders other than lumbar radiculopathy (e.g., peripheral neuropathy, multiple sclerosis).
  * Severe comorbid conditions that might interfere with the study (e.g., uncontrolled diabetes, severe cardiovascular disease).
  * Pregnant or breastfeeding women.
  * Participation in another clinical trial within the last 30 days.
  * Use of medications that could affect muscle function (e.g., corticosteroids, muscle relaxants).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population includes adult patients diagnosed with chronic lumbar radiculopathy, experiencing persistent lower back pain and/or radiating leg pain. Participants are selected from outpatient clinics and must meet specific inclusion criteria, such as the absence of recent lower limb injuries or surgeries.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Comparison of Muscle Contraction Time (Tc) Between Right and Left Gastrocnemius Muscles in Patients with Chronic Lumbar Radiculopathy | At baseline (single session)" This fits well if you're measuring contraction times of the gastrocnemius muscles in one session.
  This outcome measures the difference in muscle contraction time (Tc) between the right and left gastrocnemius muscles in patients diagnosed with chronic lumbar radiculopathy. Muscle contraction time is assessed using tensiomyography (TMG)

CONTACTS AND LOCATIONS:
Locations (1):
- Cleopatra October Hospital, Sixth of October, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tous-Fajardo J, Moras G, Rodriguez-Jimenez S, Usach R, Doutres DM, Maffiuletti NA. Inter-rater reliability of muscle contractile property measurements using non-invasive tensiomyography. J Electromyogr Kinesiol. 2010 Aug;20(4):761-6. doi: 10.1016/j.jelekin.2010.02.008. Epub 2010 Mar 16. PMID 20236839
- [Background] Schmid AB, Fundaun J, Tampin B. Entrapment neuropathies: a contemporary approach to pathophysiology, clinical assessment, and management. Pain Rep. 2020 Jul 22;5(4):e829. doi: 10.1097/PR9.0000000000000829. eCollection 2020 Jul-Aug. PMID 32766466